CLINICAL TRIAL: NCT01109069
Title: A Long-term Safety Study of Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in B Cell Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: Safety and Tolerability Study of PCI-32765 in B Cell Lymphoma and Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1103-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Diffuse Well-differentiated Lymphocytic Lymphoma; B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; B-Cell Diffuse Lymphoma
Keywords: PCI-32765; Lymphoma, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell; Bruton's Tyrosine Kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Leukemia, Lymphoid; Leukemia, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 (Experimental)
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — Dose based on parent protocol

SUMMARY:
The purpose of this study is to determine the long-term safety of a fixed-dose, daily regimen of PCI-32765 PO in subjects with B cell lymphoma or chronic lymphocytic leukemia/small lymphocytic leukemia (CLL/SLL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with recurrent surface immunoglobulin positive B cell non-Hodgkin's lymphoma (NHL) according to WHO classification (including, but not limited to, CLL/SLL, Waldenström's macroglobulinemia [WM], mantle cell lymphoma [MCL], and diffuse large B cell lymphoma [DLBCL) who have met requirements for roll over from their parent protocol and want to continue study drug.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 3 days of the first dose of study drug and agree to use dual methods of contraception during the study and for 1 month following the last dose with study drug. Post menopausal females (>45 years old and without menses for >1 year) and surgically sterilized females are exempt from this criterion.
* Male subjects must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
* Known history of Human Immunodeficiency Virus (HIV) or active infection with Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) or any uncontrolled active systemic infection.
* Lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-06; Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Dean, MD, Study Director — Medical Monitor
Locations (16):
- United States (16):
  - Stanford University, Stanford, California
  - Stanford, California
  - University of Chicago, Chicago, Illinois
  - Boston, Massachusetts
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Columbus, Ohio
  - Springfield, Oregon
  - Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Houston, Texas
  - Tyler, Texas
  - Fletcher Allen Health Care and University of Vermont, Burlington, Vermont
  - Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum K, Sharman JP, Wierda W, Zhao W, Heerema NA, Luan Y, Liu EA, Dean JP, O'Brien S. Ibrutinib Treatment for First-Line and Relapsed/Refractory Chronic Lymphocytic Leukemia: Final Analysis of the Pivotal Phase Ib/II PCYC-1102 Study. Clin Cancer Res. 2020 Aug 1;26(15):3918-3927. doi: 10.1158/1078-0432.CCR-19-2856. Epub 2020 Mar 24. PMID 32209572
- [Derived] Coutre SE, Byrd JC, Hillmen P, Barrientos JC, Barr PM, Devereux S, Robak T, Kipps TJ, Schuh A, Moreno C, Furman RR, Burger JA, O'Dwyer M, Ghia P, Valentino R, Chang S, Dean JP, James DF, O'Brien SM. Long-term safety of single-agent ibrutinib in patients with chronic lymphocytic leukemia in 3 pivotal studies. Blood Adv. 2019 Jun 25;3(12):1799-1807. doi: 10.1182/bloodadvances.2018028761. PMID 31196847
- [Derived] O'Brien S, Furman RR, Coutre S, Flinn IW, Burger JA, Blum K, Sharman J, Wierda W, Jones J, Zhao W, Heerema NA, Johnson AJ, Luan Y, James DF, Chu AD, Byrd JC. Single-agent ibrutinib in treatment-naive and relapsed/refractory chronic lymphocytic leukemia: a 5-year experience. Blood. 2018 Apr 26;131(17):1910-1919. doi: 10.1182/blood-2017-10-810044. Epub 2018 Feb 2. PMID 29437592
- See also: Home page of Pharmacyclics — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 July 2010 (the first Patient enrolled) to 31 March 2016 (the Last patient enrolled), Study was approved on June 2010.
Pre-assignment Details: This study was open to subjects from prior ibrutinib studies who met eligibility criteria for rollover from their parent study and wanted to continue receiving study drug.
Groups:
- A LONG-TERM SAFETY STUDY OF BRUTON'S TYROSINE KINASE (BTK) INH: A Long-term Safety Study of Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in B Cell Lymphoma and Chronic Lymphocytic Leukemia. This is a multicenter(16 sites in the USA), open-label, monotherapy, long-term extension study designed to evaluate the long-term (> 6 months) safety and tolerability of a fixed daily dosing regimen of ibrutinib. Ibrutinib was supplied as 140 mg or 40 mg capsules for oral administration. Subjects were to receive daily administration of a fixed dose of ibrutinib at the same dose level as in the parent study (up to 840 mg).
Period: Overall Study
Arm/Group | A LONG-TERM SAFETY STUDY OF BRUTON'S TYROSINE KINASE (BTK) INH
Started | 199
Completed | 106
Not Completed | 93

BASELINE CHARACTERISTICS:
Population: A total of 199 subjects were enrolled and received at least 1 dose of study treatment and therefore comprised the safety population which was used for safety analyses.
Arm/Group | A Long-term Safety Study of Bruton's Tyrosine Kinase (Btk) Inh
Number analyzed (Participants) | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 83
  >=65 years | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 192
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 185
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 199
Estimated creatinine clearance rate (mL/min) [Mean (Standard Deviation); unit: ML/min] | 85.55 (34.150)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Subjects were to receive ibrutinib once daily at the dose level the subject was receiving in the parent study until disease progression or unacceptable toxicity. The study included Screening, Treatment (from the first dose until study drug discontinuation), and Follow-up Phases.
Time Frame: 30 days after last dose of study drug, continue up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | A LONG-TERM SAFETY STUDY OF BRUTON'S TYROSINE KINASE (BTK) INH
Number analyzed (Participants) | 199
Participants | 199

2. Secondary Outcome: Progressive Disease (PD)
Description: A progressive disease confirmed by a CT scan.
Time Frame: 30 days after last dose of study drug, continue up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- IBRUTINIB/PCI-32765: This was a multicenter, open-label, monotherapy, long-term extension study designed to evaluate the long-term (> 6 months) safety and tolerability of a fixed daily dosing regimen of ibrutinib. PCI-32765: Dose based on parent protocol CLL: chronic lymphocytic leukemia/ SLL: small lymphocytic lymphoma.
Arm/Group | IBRUTINIB/PCI-32765
Number analyzed (Participants) | 199
Participants | 70

3. Secondary Outcome: Death Event
Description: All death events are due to AE, progressive disease, and other reasons.
Time Frame: 30 days after last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | IBRUTINIB/PCI-32765
Number analyzed (Participants) | 199
Participants | 42

4. Secondary Outcome: Documented Responses
Description: Investigator-assessed responses were summarized descriptively for subjects with CLL/SLL and listed for subjects with other NHLs based on the efficacy population.
Time Frame: 30 days after last dose of study drug, continue up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | IBRUTINIB/PCI-32765
Number analyzed (Participants) | 199
Participants
  CLL/SLL | 180
  Other NHL | 16
  Treatment discontinuation | 3

ADVERSE EVENTS:
Time Frame: 8 Years, 5 months. This is a safety longterm follow-up study, it doesn't have any common milestones.
Description: Adverse event data collection included Grade 3 or 4 AEs and major hemorrhage AEs, and the following: Grade 2 or higher eye-related AEs, and AEs of any grade that were serious, an +other malignancy, or led to dose reduction or treatment discontinuation.
Arm/Group | IBRUTINIB/PCI-32765
All-Cause Mortality (participants affected / at risk) | 111/199
Serious Adverse Events (participants affected / at risk) | 111/199
Other Adverse Events (participants affected / at risk) | 114/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBRUTINIB/PCI-32765 (N=199)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 21 (25)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Subendocardial ischaemia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Haematotympanum (Ear and labyrinth disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 8 (9)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 32 (61)
Cellulitis (Infections and infestations) | 13 (16)
Sepsis (Infections and infestations) | 11 (12)
Urinary tract infection (Infections and infestations) | 6 (7)
Gastroenteritis (Infections and infestations) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 3 (4)
Herpes zoster (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (3)
Gastroenteritis clostridial (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (3)
Localised infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 2 (3)
Urosepsis (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Clostridial sepsis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Fusarium infection (Infections and infestations) | 1 (3)
Gangrene (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Autoimmune neuropathy (Nervous system disorders) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (4)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBRUTINIB/PCI-32765 (N=199)
Neutropenia (Blood and lymphatic system disorders) | 21 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (23)
Cataract (Ear and labyrinth disorders) | 14 (20)
Diarrohea (Gastrointestinal disorders) | 9 (10)
Upper Respiratory Track Infection (Infections and infestations) | 9 (10)
Lymphocyte count decreased (Investigations) | 24 (59)
Neutrophil Count decreased (Investigations) | 17 (32)
White Blood cell count decreased (Investigations) | 8 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (15)
Hypertension (Vascular disorders) | 67 (197)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of the study are submitted for publication (ii) notification that submission of the multicenter results is no longer planned (iii) 18 months after study termination.

DOCUMENTS (1):
  • Study Protocol (2015-05-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT01109069/Prot_000.pdf